CLINICAL TRIAL: NCT05039125
Title: Comparison Between The Effects Of Different Frequencies Of Ultrasonic Cavitation On Abdominal Adiposity And Female Hormones In Polycystic Ovarian Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 62
Record Dates: First submitted 2021-09-01; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 40000HZ ultrasound cavitation (Active Comparator): group A (n=15) received 40000HZ ultrasound cavitation, Treatment time was 30 minutes /sessions, 3 times/ week for two months. Both groups (A and B) received a low caloric diet (1200 Kcal/day). All participants had their medical treatment as prescribed by the physician.
  Interventions: Radiation: ultrasonic cavitation
- 2600HZ ultrasound cavitation (Active Comparator): group B (n=15) received 2600HZ ultrasound cavitation. Treatment time was 30 minutes /sessions, 3 times/ week for two months. Both groups (A and B) received a low caloric diet (1200 Kcal/day). All participants had their medical treatment as prescribed by the physician.
  Interventions: Radiation: ultrasonic cavitation

INTERVENTIONS:
Radiation: ultrasonic cavitation — * From a standing position, each participant's abdomen was divided transversally into three sections; resulting in a total of 6 abdominal segments.
  * Part III: 3cm above the umbilicus to 2cm below the umbilicus
  * After washing the skin on the anterior abdominal wall with alcohol, a conducting medium (gel) was placed to the ultrasonic instrument's cavitational head.
  * The gadget was turned on, a 30-minute timer was set, and the intensity was gradually increased.
  * The cavitation head then moved extremely gently in a small circular motion on each abdomen section for 5 minutes.
  * After completing the ultrasonic application to the six regions of the abdomen, the skin was cleansed with a piece of cotton.
  For group (A): 40000 HZ ultrasound was delivered for 30 minutes, 3 times/week for 2 months.
  For group (B):26000 HZ ultrasound was delivered for 30 minutes, 3 times/week for 2 months

SUMMARY:
Thirty women diagnosed with PCOS had participated in the study. They suffered from amenorrhea or oligo-menorrhea and subcapsular follicles. Their ages were from 20-35 years. Their BMI was from 30 - 35 kg/m². Their waist/hip ratio was ˃ 0.85. Their LH/FSH ratio was ≥ 1.5. They were recruited randomly from the outpatient clinic of gynecology in Minya governorate hospital. They were randomly assigned into two groups equal in number: (A and B); group A (n=15) received 40000HZ ultrasound cavitation, group B (n=15) received 2600HZ ultrasound cavitation. Treatment time was 30 minutes /sessions, 3 times/ week for two months. Both groups (A and B) received a low caloric diet (1200 Kcal/day). All participants had their medical treatment as prescribed by the physician.

DETAILED DESCRIPTION:
Participants in both groups were told to follow a low calorie diet (1200 Kcal/day) tailored to their specific needs (low in fat (15%), high in complex carbs (55%), and adequate in protein) (30 percent ) (11).

The application procedure of ultrasound cavitation for both groups (A and B):-

* Each participant in both groups (A and B) received instructions on the treatment techniques as well as the benefits of the USFC.
* To improve lymphatic drainage, each subject was encouraged to consume one liter of water before and after the therapy sessions.
* Each participant was urged to empty her bladder before beginning each treatment session so order to remain comfortable and relaxed throughout the session.
* From a standing position, each participant's abdomen was divided transversally into three sections; see fig (1) 1- Part I: from the xiphoid process to 3cm above the umbilicus, 2- Section II: from 2cm below the umbilicus to the pubic bone, and vertically to the linea alba, each part was separated into right and left segments, resulting in a total of 6 abdominal segments.
* Part III: 3cm above the umbilicus to 2cm below the umbilicus
* After washing the skin on the anterior abdominal wall with alcohol, a conducting medium (gel) was placed to the ultrasonic instrument's cavitational head.
* The gadget was turned on, a 30-minute timer was set, and the intensity was gradually increased.
* The cavitation head then moved extremely gently in a small circular motion on each abdomen section for 5 minutes.
* After completing the ultrasonic application to the six regions of the abdomen, the skin was cleansed with a piece of cotton.

For group (A): 40000 HZ ultrasound was delivered for 30 minutes, 3 times/week for 2 months.

For group (B):26000 HZ ultrasound was delivered for 30 minutes, 3 times/week for 2 months

ELIGIBILITY:
Inclusion Criteria:

* nulligravida women with PCOS complaining of at least one year of infertility. They suffered from amenorrhea or oligo-menorrhea and subcapsular follicles. Their ages ranged from 20-35 years. Their BMI ranged from 30-35 kg/m². Their waist/hip ratio was ˃ 0.85. Their LH/FSH ratio was ≥ 1.5. They were from the same social class.

Exclusion Criteria:

* history of heart disease, high cholesterol, l iver or kidney diseases, diabetes mellitus, hypertension, pregnancy, scarring, hernias, or skin diseases in the abdominal region that prevent the application of ultrasound cavitation

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Anthropometric measures | 2 moths after treatment
  Weight-Height scale was used for each participant of the two studied groups (A & B) before and after the study to measure the weight and height

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed Maged M ElGoly, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No